CLINICAL TRIAL: NCT06441851
Title: Randomized Clinical Trial to Compare Two Partial Nephrectomy Techniques for Renal Tumors: Robot-assisted vs Videolaparoscopic
Brief Title: Study to Compare Two Partial Nephrectomy Techniques for Renal Tumors: Robot-assisted vs Videolaparoscopic
Acronym: VPN x RANP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, MAURICIO DENER CORDEIRO, Principal Investigator, MD, PhD, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP5030/2023
Record Dates: First submitted 2024-04-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Renal Cancer
Keywords: Renal cancer; Nephrectomy; Partial nephrectomy; Videolaparoscopic partial nephrectomy; Robot-assisted partial nephrectomy
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaparoscopic Partial Nephrectomy (VPN) (Active Comparator): Patients randomized to VPN group will be submitted to a videolaparoscopic partial nephrectomy in which lesion will be identified, renal artery will be selectively clamped and renal parenchyma will be section with scissors and cautery. Suture will be made in two planes with absorbable sutures.
  Interventions: Procedure: Videolaparoscopic Partial Nephrectomy
- Robot-assisted Partial Nephrectomy (RANP) (Experimental): Patients randomized to RAN'P group will be submitted to a robot-assisted partial nephrectomy in which lesion will be identified, renal artery will be selectively clamped and renal parenchyma will be section with scissors and cautery. Suture will be made in two planes with absorbable sutures.
  Interventions: Procedure: Robot-assisted Partial Nephrectomy

INTERVENTIONS:
Procedure: Videolaparoscopic Partial Nephrectomy — Videolaparoscopic partial nephrectomy
  Other Names: VPN
  Arms: Videolaparoscopic Partial Nephrectomy (VPN)
Procedure: Robot-assisted Partial Nephrectomy — Robot-assisted partial nephrectomy
  Other Names: RAPN
  Arms: Robot-assisted Partial Nephrectomy (RANP)

SUMMARY:
Randomized, open-label clinical trial to compare renal volumetry pre and post operative in patients undergoing two types of partial nephrectomy techniques for renal tumors: robot-assisted vs videolaparoscopic.

DETAILED DESCRIPTION:
Renal tumors are an important public health issue, representing approximately 4,2% of all newly diagnosed cancers around the world. Renal tumors are more prevalent in adults over 45 years old, and with higher frequency in men than women. Many risks factor have already been identified, including smoking (increase in twice the renal cancer risk), obesity, hypertension, and renal cancer familiar history.

Surgery is one of the main treatment options for renal tumors and is considered the only curative treatment for localized ones. The most common surgeries used to treat it are Partial Nephrectomy (PN) and Radical Nephrectomy (RN). PN in indicated for smaller tumors (smaller than 4cm size) once it has already demonstrated renal function preservation and decrease chronic kidney disease (CDK) risk and cardiovascular events. Furthermore, RN is indicated for bigger tumors or for those who are centrally located in the middle of the kidney.

In the last years, PN use have been increased and consequently, RN use has been decreased.

According to a recent published study, PN use for T1a tumors increased from 20,2% in 2004, to 59,7% in 2015. Furthermore, 5-year cancer survival rates between patients undergone PN or RN was similar, with PN being more associated with lower general mortality rates. However, PN is technically more challenging and is associated with complications and local higher recurrence risks.

Both are viable surgery options for renal tumors and the chosen technique of them should be considered according to surgeon expertise, patient's comorbidities, and tumor characteristics.

There are some PN ways, including Open (OPN), Laparoscopic (LPN) and robot-assisted (RAPN), however the best technique is still unknown. Some studies have been comparing this three, and a recent 39-studies metanalysis evaluating 11.310 patients reported RAPN is which presented lower general complications, less warm ischemia period, and higher kidney function preservation rates in comparison with LPN or OPN. Other 29-studies metanalysis evaluating 5952 patients showed RAPN presented lower surgical and hospitalization periods compared to OPN and LPN. However, RANP is associated with higher costs and a longer learning curve than other NP techniques.

Renal volumetry is an important measure for kidney function evaluation which aids on surgical approach choose for NP. In the present, there are some ways to evaluate pre and post operative kidney volumetry such as TC, RMN, and 3D ultrasonography (3DUS). A systematic review and metanalysis of 26 studies analyzed 1918 patients, and showed TC preoperative renal volumetry is the best way to predict postoperative kidney function and the need for a NP. Renal volumetry by TC and RMN postoperative also were considered good trustful measures to evaluate volumetry and remained kidney functions after PN. 3DUS appear to be a more economic and good measure to evaluate it with a good precision compared to what was found to TC and RMN.

In general, pre and postoperative renal volumetry are an important measure to guide surgeons on the best surgery approach in PN, and right renal volumetry image evaluation should be considered according to costs available, patients characteristics and surgeon experience. Then, this study aims to compare NP techniques (VPN and RAPN) using renal volumetry pre and postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 99 years old;
* Patients with non-metastatic renal cancer (confirmed by pre operatory TC);
* Patients eligible for videolaparoscopic partial nephrectomy;
* Patients who signed study informed consent form

Exclusion Criteria:

* Pregnant patients;
* Patients with concomitant indications with nephrectomy;
* Patients with a clinical condition that contraindicates nephrectomy;
* Patients with a clinical condition that contraindicates robot-assisted surgeries (determined by urology team);
* Patients with previous surgeries that contraindicates robot-assisted surgeries (determined by urology team);

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Renal volumetry | Up to 6 months after surgery
  Renal volumetry measured by computadorized tomography

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell S, Uzzo RG, Allaf ME, Bass EB, Cadeddu JA, Chang A, Clark PE, Davis BJ, Derweesh IH, Giambarresi L, Gervais DA, Hu SL, Lane BR, Leibovich BC, Pierorazio PM. Renal Mass and Localized Renal Cancer: AUA Guideline. J Urol. 2017 Sep;198(3):520-529. doi: 10.1016/j.juro.2017.04.100. Epub 2017 May 4. PMID 28479239
- [Background] Kutikov A, Uzzo RG. The R.E.N.A.L. nephrometry score: a comprehensive standardized system for quantitating renal tumor size, location and depth. J Urol. 2009 Sep;182(3):844-53. doi: 10.1016/j.juro.2009.05.035. Epub 2009 Jul 17. PMID 19616235
- [Background] Thompson RH, Lane BR, Lohse CM, Leibovich BC, Fergany A, Frank I, Gill IS, Blute ML, Campbell SC. Every minute counts when the renal hilum is clamped during partial nephrectomy. Eur Urol. 2010 Sep;58(3):340-5. doi: 10.1016/j.eururo.2010.05.047. Epub 2010 Jun 9. PMID 20825756
- [Background] Kim SP, Thompson RH, Boorjian SA, Weight CJ, Han LC, Murad MH, Shippee ND, Erwin PJ, Costello BA, Chow GK, Leibovich BC. Comparative effectiveness for survival and renal function of partial and radical nephrectomy for localized renal tumors: a systematic review and meta-analysis. J Urol. 2012 Jul;188(1):51-7. doi: 10.1016/j.juro.2012.03.006. Epub 2012 May 14. PMID 22591957
- [Background] Kutikov A, Egleston BL, Canter D, Smaldone MC, Wong YN, Uzzo RG. Competing risks of death in patients with localized renal cell carcinoma: a comorbidity based model. J Urol. 2012 Dec;188(6):2077-83. doi: 10.1016/j.juro.2012.07.100. Epub 2012 Oct 18. PMID 23083850
- [Background] Venkatesan AM, Kundu S, Sacks D, Wallace MJ, Wojak JC, Rose SC, Clark TW, d'Othee BJ, Itkin M, Jones RS, Miller DL, Owens CA, Rajan DK, Stokes LS, Swan TL, Towbin RB, Cardella JF; Society of Interventional Radiology Standards of Practice Committee. Practice guidelines for adult antibiotic prophylaxis during vascular and interventional radiology procedures. Written by the Standards of Practice Committee for the Society of Interventional Radiology and Endorsed by the Cardiovascular Interventional Radiological Society of Europe and Canadian Interventional Radiology Association [corrected]. J Vasc Interv Radiol. 2010 Nov;21(11):1611-30; quiz 1631. doi: 10.1016/j.jvir.2010.07.018. No abstract available. PMID 21029949
- [Background] Lane BR, Abouassaly R, Gao T, Weight CJ, Hernandez AV, Larson BT, Kaouk JH, Gill IS, Campbell SC. Active treatment of localized renal tumors may not impact overall survival in patients aged 75 years or older. Cancer. 2010 Jul 1;116(13):3119-26. doi: 10.1002/cncr.25184. PMID 20564627
- [Background] Zini L, Perrotte P, Capitanio U, Jeldres C, Shariat SF, Antebi E, Saad F, Patard JJ, Montorsi F, Karakiewicz PI. Radical versus partial nephrectomy: effect on overall and noncancer mortality. Cancer. 2009 Apr 1;115(7):1465-71. doi: 10.1002/cncr.24035. PMID 19195042
- [Background] Ficarra V, Novara G, Secco S, Macchi V, Porzionato A, De Caro R, Artibani W. Preoperative aspects and dimensions used for an anatomical (PADUA) classification of renal tumours in patients who are candidates for nephron-sparing surgery. Eur Urol. 2009 Nov;56(5):786-93. doi: 10.1016/j.eururo.2009.07.040. Epub 2009 Aug 4. PMID 19665284